CLINICAL TRIAL: NCT00531518
Title: Early Detection and Intervention for the Prevention of Psychosis Project
Brief Title: Early Detection and Intervention for the Prevention of Psychosis
Acronym: EDIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, William McFarlane, Principal Investigator, MaineHealth
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 58920; RWJF #58920 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia; Bipolar Disorder; Depression; Psychotic Disorders
Keywords: Schizophrenia; Bipolar disorder; Psychosis; Prodromal psychosis; Family psychoeducation; Supported education; Supported employment; Ulra-high-risk for psychosis; Major depression; Bipolar disorder, with psychotic features; Major depression, with psychotic features; Attenuated, prodromal psychotic symptoms
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depression; Psychotic Disorders; Depressive Disorder, Major | interventions — Aripiprazole; Fluoxetine; Bupropion; Sertraline; Lamotrigine; Psychotherapy, Group; Employment, Supported; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): This is the control arm. Participants will be offered only case management. Participants may seek outside treatment, without guidance from study staff.
- Family-aided Assertive Community Treatment (Experimental): This is the experimental intervention arm for high-risk-for-psychosis participants. The intervention includes psychiatric drugs (aripiprazole; fluoxetine; bupropion; sertraline; lamotrigine), psychoeducational multifamily group treatment and supported employment and education .
  Interventions: Drug: aripiprazole; fluoxetine; bupropion; sertraline; lamotrigine; Behavioral: Psychoeducational multifamily group treatment; Behavioral: Supported employment and education

INTERVENTIONS:
Drug: aripiprazole; fluoxetine; bupropion; sertraline; lamotrigine — Oral, daily, generally at lower than manufacturer's recommendations
  Other Names: Abilify; Prozac; Welbutrin; Zoloft; Lamictal
  Arms: Family-aided Assertive Community Treatment
Behavioral: Psychoeducational multifamily group treatment — Families and patients are educated on psychobiology of psychosis and trained in coping skills to avoid psychosis by reducing stress and optimizing social environment at home, school, work
  Other Names: Family psychoeducation,; Family behavioral therapy; Multiple family group therapy
  Arms: Family-aided Assertive Community Treatment
Behavioral: Supported employment and education — Participants are provided direct assistance, guidance and ongoing support to gain employment and succeed in their educational goals.
  Other Names: Supported employment; Supported education
  Arms: Family-aided Assertive Community Treatment

SUMMARY:
EDIPP is a multisite trial of early identification and intervention to prevent the onset of psychosis in adolescents and young adults, carried out at six sites across the United States. The hypothesis is that very early identification and intervention will be effective in delaying or preventing onset of psychosis and improving social and occupational functioning.

DETAILED DESCRIPTION:
The study is structured as a cutoff, regression discontinuity design, in which lower risk-for-psychosis participants will not be treated by protocol but followed up for two years. Those at higher risk will be treated with anti-psychotic, antidepressant and mood stabilizing medications by symptom indications, and systematically provided psychoeducational multifamily group treatment, supported education and employment, and intensive clinical case management, using key elements of Assertive Community Treatment. Both arms of the study will be followed for two years and assessed at 6, 12, and 24 months. Outcome measures include rates of conversion to psychosis, relapse of psychosis, development of psychotic disorder diagnoses, levels of positive, negative and general symptoms, social and vocational functioning, family functioning, and neurocognitive functioning.

The six sites include Sacramento, California; Salem Oregon; and surrounding counties, Ypsilanti and Washtenaw County, Michigan; Portland, Maine; Albuquerque, New Mexico and Glen Oaks, New York.

In addition to symptomatic and functional outcomes, impact on incidence of psychotic disorders, including schizophrenia, will be assessed, as will cost-benefit effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the age range of 12-25 and living in the experimental catchment area may be enrolled in the EDIPP study based on meeting at least one of the inclusion requirements AND none of the exclusion criteria;
* Screening process indicates symptoms equivalent to a minimum rating of '1' on at least one positive symptom of psychosis;
* Screening process indicates a likely family history of first degree relative with psychotic illness plus a deterioration in functioning equivalent to a 30% drop in functioning score over the past year; OR
* Screening process indicates a likely history of schizotypal personality disorder plus a deterioration in functioning equivalent to a 30% drop in functioning over the past year.

Exclusion Criteria:

* Outside the age range of 12 to 25 years;
* History of intelligence quotient (IQ) below 70 (based on school records, not tested at PIER);
* More than one month duration of psychosis (guided by the criteria of at least one 6 on the Positive Symptom sub-scale of the Scale of Positive Symptoms (SOPS);
* History of previous psychotic episode, whether or not treatment was received;
* Taken antipsychotic medication for more than 30 days at a therapeutic dose for psychotic symptoms;
* Either the young person being screened for the study or both parents do not speak proficient English;
* Female is pregnant at baseline (inquired on the screening interview); AND
* Subject is a prisoner.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 292 (Actual)
Dates: Start 2007-10; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R. McFarlane, M.D., Principal Investigator — MaineHealth
Locations (6):
- United States (6):
  - University of California-Davis, Imaging Research Center, Sacramento, California
  - Portland Identification and Early Referral Program, Portland, Maine
  - Washtenaw County, Ann Arbor, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Zucker Hillside Hosptial, Glen Oaks, New York
  - Mid-Valley Behavioral Care Network, Salem, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Currently, on request, data will be shared with legitimate organizations for specific analyses approved by the PI and the Maine Medical Center Institutional Review Board.

REFERENCES:
- [Result] Lynch S, McFarlane WR, Joly B, Adelsheim S, Auther A, Cornblatt BA, Migliorati M, Ragland JD, Sale T, Spring E, Calkins R, Carter CS, Jaynes R, Taylor SF, Downing D. Early Detection, Intervention and Prevention of Psychosis Program: Community Outreach and Early Identification at Six U.S. Sites. Psychiatr Serv. 2016 May 1;67(5):510-6. doi: 10.1176/appi.ps.201300236. Epub 2016 Jan 14. PMID 26766751
- [Result] McFarlane WR, Levin B, Travis L, Lucas FL, Lynch S, Verdi M, Williams D, Adelsheim S, Calkins R, Carter CS, Cornblatt B, Taylor SF, Auther AM, McFarland B, Melton R, Migliorati M, Niendam T, Ragland JD, Sale T, Salvador M, Spring E. Clinical and functional outcomes after 2 years in the early detection and intervention for the prevention of psychosis multisite effectiveness trial. Schizophr Bull. 2015 Jan;41(1):30-43. doi: 10.1093/schbul/sbu108. Epub 2014 Jul 26. PMID 25065017
- See also: Describes the orientation of the program and early signs of psychosis — http://www.preventmentalillness.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Family-aided Assertive Community Treatment
Started | 87 | 205
Completed | 55 | 134
Not Completed | 32 | 71

BASELINE CHARACTERISTICS:
Population: All eligible participants (n=292) were entered into the outcome analysis. This was an intent-to-treat study and statistical analysis.
Groups:
- Experimental Intervention: This is the experimental intervention arm for high-risk-for-psychosis participants. The intervention includes psychiatric drugs (aripiprazole; fluoxetine; bupropion; sertraline; lamotrigine), psychoeducational multifamily group treatment and supported employment and education .
  aripiprazole; fluoxetine; bupropion; sertraline; lamotrigine: Oral, daily, generally at lower than manufacturer's recommendations
  Psychoeducational multifamily group treatment: Families and patients are educated on psychobiology of psychosis and trained in coping skills to avoid psychosis by reducing stress and optimizing social environment at home, school, work
  Supported employment and education: Participants are provided direct assistance, guidance and ongoing support to gain employment and succeed in their educational goals.
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Intervention | Total
Number analyzed (Participants) | 87 | 205 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.23 (3.18) | 16.40 (3.30) | 16.35 (3.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 89 | 115
  Male | 61 | 116 | 177
Region of Enrollment [Number; unit: participants]
  United States | 87 | 205 | 292
Psychotic symptoms [Mean (Standard Deviation); unit: units on a scale] — Psychotic symptoms were assessed and scored using the Structured Interview for the Prodromal Syndrome (SIPS) and the Scale of Prodromal Symptoms (SOPS). The SOPS provides a measure of four domains of symptoms, including positive, negative, disorganized and general symptoms. The Positive Symptom sub-scale score reported is the sum of all five symptom items in the Positive Symptom sub-scale. The Positive Symptom sub-scale assesses psychotic symptoms, each item on a scale of 0-6. The sum scale score is 0-30, with 30 indicating severe psychotic symptoms, while 0 indicates no psychotic symptoms.
  units on a scale | 4.15 (1.76) | 11.99 (3.42) | 9.65 (4.69)

OUTCOME MEASURES:

1. Primary Outcome: Psychotic Symptoms
Description: Psychotic symptoms were assessed and scored using the Structured Interview for the Prodromal Syndrome (SIPS) and the Scale of Prodromal Symptoms (SOPS). The SOPS provides a measure of four domains of symptoms, including positive, negative, disorganized and general symptoms. The Positive Symptom sub-scale score reported is the sum of all five symptom items in the Positive Symptom sub-scale. The Positive Symptom sub-scale assesses psychotic symptoms, each item on a scale of 0-6. The sum scale score is 0-30, with 30 indicating severe psychotic symptoms, while 0 indicates no psychotic symptoms.
Time Frame: two years
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: This is the control arm. Participants will be offered only case management. Participants may seek outside treatment, without guidance from study staff.
Arm/Group | Control | Family-aided Assertive Community Treatment
Number analyzed (Participants) | 87 | 205
units on a scale | 9.2 (1.0) | 6.7 (0.4)
Statistical Analysis 1: Comparison: Control vs Family-aided Assertive Community Treatment; The analysis used regression discontinuity methods, in which the baseline sum scores were adjusted and centered to an equalize control and experimental conditions; Test type: Superiority or Other; p = .0034, Mixed Models Analysis — The final analysis included adjstment for site and baseline sum psychotic symptom score

ADVERSE EVENTS:
Time Frame: Over 24 months
Arm/Group | Control Group | Family-aided Assertive Community Treatment
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/205
Other Adverse Events (participants affected / at risk) | 19/87 | 51/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=87) | Family-aided Assertive Community Treatment (N=205)
suicide (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=87) | Family-aided Assertive Community Treatment (N=205)
Negative events (Psychiatric disorders) | 19 (19) | 51 (51) — "Negative events" is the measure that includes hospitalizations, incarcerations, assaults, suicides and suicide attempts. It is the sum of such events within each experimental treatment condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No